CLINICAL TRIAL: NCT06125041
Title: A Single-arm, Multi-center and Exploratory Study of Adebelizumab Combined With Chemotherapy and Sequential Adebelizumab Combined With Radiotherapy in the Treatment of Newly Diagnosed Extensive Small Cell Lung Cancer
Brief Title: Adebelizumab Combined With Chemotherapy and Radiotherapy Treat ES-SCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Jiandong Zhang, Director of radiotherapy department,archiater, Qianfoshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YXLL-KY-2023(102)
Record Dates: First submitted 2023-09-18; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Extensive Small Cell Lung Cancer
MeSH Terms: interventions — Drug Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Administration regimen: adebelizumab 1200mg, IV, Q3W+ carboplatin AUC 5 d1+ etoposide 100mg/m2 D1, 2, 3; 21 days is a treatment cycle. After 4-6 cycles, patients with imaging evaluation CR/PR/SD (according to tumor RECIST1.1 standard) receive adebelizumab maintenance therapy and radiotherapy at the same time. Patients with imaging evaluation PD (according to tumor RECIST1.1 standard) can receive adebelizumab maintenance therapy combined with radiotherapy according to the clinical practice, or they can change other treatment schemes and continue to follow up.
  After the induction treatment, the participants will continue to receive adebelizumab (20mg/kg, IV, Q3W) combined with concurrent radiotherapy (conventional radiotherapy SBRT chest lesions (2Gy*25f), brain (3Gy*10f)/ bone (3Gy*10f)/ suprarenal gland (3Gy*10-15f)/ liver (3YX).
  Interventions: Drug: Adebelizumab+Carboplatin+Etoposide+Concurrent Radiotherapy

INTERVENTIONS:
Drug: Adebelizumab+Carboplatin+Etoposide+Concurrent Radiotherapy — Eligible patients will receive the following treatment schemes: adebelizumab+carboplatin+etoposide, with one treatment cycle every three weeks. After 4-6 cycles, adebelizumab maintenance therapy combined with concurrent radiotherapy will be given, and conventional radiotherapy will be given to chest lesions (2Gy*(20-30)f), brain (3Gy*10f)/ bone (3Gy*10f)/ adrenal gland. Immunotherapy is suspended during radiotherapy for chest lesions and lymph nodes in mediastinum, and immunotherapy is given 1-2 weeks after radiotherapy. Radiotherapy for other metastatic lesions can be carried out simultaneously with immunotherapy.
  Other Names: Adebelizumab Combined With Chemotherapy and Sequential Adebelizumab Combined With Radiotherapy in the Treatment of Newly Diagnosed Extensive Small Cell Lung Cancer

SUMMARY:
To observe the efficacy and safety of adebelizumab combined with chemotherapy and sequential adebelizumab combined with radiotherapy in the treatment of newly diagnosed extensive small cell lung cancer.

DETAILED DESCRIPTION:
This study is a one-arm, multi-center and exploratory study. Eligible patients will receive the following treatment schemes: adebelizumab+carboplatin+etoposide, with one treatment cycle every three weeks. After 4-6 cycles, adebelizumab maintenance therapy combined with concurrent radiotherapy will be given, and conventional radiotherapy will be given to chest lesions (2Gy*(20-30)f), brain (3Gy*10f)/ bone (3Gy*10f)/ adrenal gland. Immunotherapy is suspended during radiotherapy for chest lesions and lymph nodes in mediastinum, and immunotherapy is given 1-2 weeks after radiotherapy. Radiotherapy for other metastatic lesions can be carried out simultaneously with immunotherapy.

Research population: patients with extensive small cell lung cancer diagnosed by histopathology or cytology, both male and female, aged 18-75 years old, who have not received systemic treatment for small cell lung cancer before. 51 patients are planned to be enrolled.

Main research end point： PFS(RECIST v1.1 standard) evaluated by researchers. Secondary end point

Key secondary study endpoints:

The incidence of adverse reactions above grade 3 in patients evaluated according to CTCAE5.0 version 5.0.

Other secondary study endpoints:

OS； ORR(RECIST v1.1 standard) evaluated by researchers; DoR； evaluated by the researcher; DCR； assessed by the researcher; PFS rate at 6 months and 1 year OS rate at 1 year and 2 years. The end point of exploratory research Explore the biomarker related to curative effect.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old, both male and female;
* Extensive small cell lung cancer (metastatic lesions ≤3 organs, ≤5 lesions) confirmed by histology or cytology (according to the Veterans Administration Lung Study Group (VALG staging), including asymptomatic brain metastasis, multiple lung metastases, supraclavicular or mediastinal lymph node metastasis, bone metastasis, adrenal metastasis, retroperitoneal lymph node metastasis, etc.;
* The score of ECOG physical condition is 0~1;
* Never received first-line systemic therapy for ES-SCLC or immune checkpoint inhibitors before;
* Previous surgical treatment did not include adjuvant therapy such as radiotherapy and chemotherapy, and there was a five-treatment interval of at least 6 months from the diagnosis of extensive SCLC to the last chemotherapy and radiotherapy.
* It is necessary to be able to provide tumor tissue samples before the experimental treatment, which can be archived within 6 months before the first dose of the research drug or freshly obtained. Specimens should be fixed in formalin and embedded in paraffin (FFPE), and at least 10 4~6μm thick sections can be cut out for staining and detection. Specimens that do not accept fine needle aspiration biopsy, cytological smears of pleural effusion drainage and centrifugation, bone lesions without soft tissue components or decalcified bone tumor specimens, and tissues drilled for biopsy are not enough for biomarker detection; Tissue samples should be submitted within 4 weeks before or after signing the notice, allowing research participants to provide Before the tumor tissue samples were taken into the study;
* Estimated survival time ≥8 weeks;
* There is a measurable lesion defined by RECIST standard v1.1: only when a previously irradiated lesion shows definite disease progression after radiotherapy and the previous lesion is not the only lesion can it be considered as a measurable lesion;
* Women of childbearing age must have a serum pregnancy study within 7 days before the first medication, and the result is negative. Participants in the study of women of childbearing age and male participants whose partners are women of childbearing age must agree to contraception within 24 weeks after signing the informed consent form to the last administration of the study drug;
* Before the first dose of study drug, the laboratory test value meets the following conditions:

  1. Blood routine (no blood transfusion and no use of hematopoietic stimulating factors within 14 days before screening) Material correction): White blood cell (WBC) ≥ 3.0× 10^9/L; Absolute neutrophil count (ANC) ≥ 1.5× 10^9/L; Platelet (PLT) ≥ 100× 10^9/L； Hemoglobin (HGB) ≥ 9.0g/dl;
  2. Liver function: aspartate aminotransferase (AST) ≤ 2.5 x ULN; Alanine aminotransferase (ALT) ≤ 2.5 x ULN, and ALT and AST≤5 x ULN； of participants in liver metastasis study; Total bilirubin (TBIL) ≤ 1.5 x ULN (except Gilbert syndrome ≤ 3.0 mg/dl);
  3. Renal function: serum creatinine ≤1.5 x ULN or creatinine clearance rate (CRCL) ≥ 50 ml/minute;
  4. Coagulation function: international normalized ratio (INR) ≤ 1.5 x ULN, activated partial thromboplastin time (APTT) ≤ 1.5 x ULN (only applicable to patients who have not received anticoagulant therapy at present, and patients who are currently receiving anticoagulant therapy should receive stable dose of anticoagulant therapy);
  5. Others: lipase ≤1.5 x ULN (if lipase > 1.5 x ULN without clinical or imaging confirmation of pancreatitis, you can be included in the group); Amylase ≤1.5 x ULN (if amylase > 1.5 x ULN without clinical or imaging confirmation of pancreatitis, you can be included in the group); Alkaline phosphatase (ALP) ≤ 2.5 ULN, and ALP ≤ 5 ULN for participants in liver metastasis or bone metastasis research.
* The study participants voluntarily joined the study, signed the informed consent, and had good compliance and cooperated with the follow-up.

Exclusion Criteria:

* Symptomatic brain metastasis and liver metastasis;
* The effusion in the third space with clinical symptoms needs repeated drainage, such as pericardial effusion, pleural effusion and peritoneal effusion that cannot be controlled by pumping or other treatments;
* Uncontrollable or symptomatic hypercalcemia;
* Other malignant tumors occurred less than 5 years before the first dose, except for cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery and ductal carcinoma in situ after radical surgery (hormone therapy for non-metastatic prostate cancer or breast cancer is allowed);
* Active, known or suspected autoimmune diseases (see Annex 4) include but are not limited to myasthenia gravis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis and inflammatory bowel disease. Allow type I diabetes (blood sugar can be controlled by insulin treatment), residual hypothyroidism caused by autoimmune thyroiditis that only needs hormone replacement therapy, or the situation that it is not expected to recur in the absence of external stimulus; In patients with eczema, psoriasis, chronic lichen simplex or only vitiligo (psoriasis arthritis should be excluded), if the skin rash coverage area is less than 10% of the body surface area, the disease has been fully controlled at baseline and only low titer is needed.
* Local steroid therapy, the basic disease did not appear acute aggravation in the past 12 months (without psoralen plus ultraviolet radiation [PUVA], methotrexate, retinoids, biological agents, oral calcineurin inhibitors, high titer or oral steroids) can enter the study;
* Previously received any T cell co-stimulation or immune checkpoint treatment, including but not limited to cytotoxic T lymphocyte associated antigen-4 (CTLA-4) inhibitor, PD-1 inhibitor, PD-L1/2 inhibitor or other drugs targeting T cells;
* Use corticosteroids (> 10 mg/day prednisone or equivalent dose) or other immunosuppressants within 14 days or less before the first dose of study drug. Inhalation or local use of steroids and adrenal glands instead of steroids is allowed without active autoimmune diseases;
* HBsAg positive and the number of copies of HBV DNA is greater than the upper limit of the normal value of the laboratory of the research center (1000 copies /ml or 500IU/ml), or HCV positive (HCV RNA or HCV Ab detection indicates acute and chronic infection); Known HIV positive history or known Acquired Immune Deficiency Syndrome (AIDS);
* Suffering from a history of idiopathic pulmonary fibrosis, organized pneumonia (such as bronchiolitis obliterans), drug-induced pneumonia, radiation pneumonia requiring steroid treatment or active pneumonia with clinical symptoms; Or other moderate or severe lung diseases that seriously affect lung function (patients with a history of radiation pneumonia (fibrosis) in the radiation area can participate in this study);
* Active pulmonary tuberculosis, TB) or research participants with a history of active pulmonary tuberculosis infection within 48 weeks or less before screening, regardless of treatment;
* There are severe infections when entering the group, including but not limited to infection complications, bacteremia, severe pneumonia, etc. that require hospitalization;
* Have undergone major surgery within 28 days before joining the group, or plan to undergo major surgery during the study period;
* Use attenuated live vaccine within 28 days before enrollment, or expect to use such attenuated live vaccine during the study period (patients are not allowed to receive attenuated live influenza vaccine within 4 weeks before randomization, during the treatment period and within 5 months after the last administration of SHR-1316/ placebo);
* Have serious cardiovascular diseases, such as heart failure of new york Heart Association (NYHA) grade 2 or above, unstable angina pectoris, unstable arrhythmia, myocardial infarction or cerebrovascular accident within the first 3 months at random;
* patients who have received allogeneic bone marrow transplantation or solid organ transplantation in the past;
* It is known to be allergic to research drugs or excipients, and it is known to have a serious allergic reaction to any kind of monoclonal antibody; Have a history of carboplatin or etoposide allergy;
* Have received any other experimental drug treatment or participated in another interventional clinical study within 4 weeks before signing ICF;
* Within one week before joining the group, he received systemic immunosuppressive drugs (including but not limited to glucocorticoid, cyclophosphamide, azathioprine, methotrexate, thalidomide and anti-tumor necrosis factor [anti -TNF] drugs). Patients receiving short-term, systemic immunosuppressant therapy, such as glucocorticoid for nausea, vomiting, or allergic reaction management or preventive medication, can be enrolled in the study with the approval of the researcher. Inhaled corticosteroids are allowed to treat patients with chronic obstructive pulmonary disease, mineralocorticoids such as hydrocortisone to treat postural hypotension, and low-dose glucocorticoid supplements to treat adrenal insufficiency;
* Known mental illness, alcoholism, inability to quit smoking, drug abuse or substance abuse; According to the judgment of the researcher, there are other factors that may lead to the forced termination of the study, such as non-compliance with the protocol, other serious diseases (including mental illness) requiring combined treatment, serious abnormal laboratory examination, family or social factors, which will affect the safety of the study participants, or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 18 month
  The time from the beginning of randomization to the occurrence (in any way) progression or death (for any reason) of a tumor.

SECONDARY OUTCOMES:
overall survival | 18 month
  Time from randomization to death (for any reason). For subjects who have been lost before death, the last follow-up time is usually calculated as the time of death.
objective response rat | 18 month
  The proportion of patients whose tumor volume has shrunk to a predetermined value and can maintain the minimum time limit is the sum of the proportion of complete remission and partial remission.
disease control rate | 18 month
  The percentage of cases with remission (PR+CR) and stable lesion (SD) after treatment to the evaluable cases.
Duration of Response | 18 month
  Refers to the first evaluation of the tumor as CR or PR.

OTHER OUTCOMES:
Explore biomarker related to curative effect | 18 month
  To explore the progression-free survival (PFS) and overall survival (OS) of patients with different types (SCLC-A/N/Y/P) of extensive small cell lung cancer treated by adebelizumab combined with chemotherapy and sequential adebelizumab combined with radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jiandong Zhang, Principal Investigator — Shandong First Medical University
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China